CLINICAL TRIAL: NCT05200312
Title: A Phase II Study of the Bruton's Tyrosine Kinase Inhibitor, Zanubrutinib, in Combination With Lenalidomide Plus Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma
Brief Title: A Phase II Study of Zanubrutinib, Lenalidomide Plus R-CHOP as the First-line Treatment for Diffused Large B-cell Lymphoma
Acronym: ZR2-CHOP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWCLL-003
Record Dates: First submitted 2022-01-17; First posted 2022-01-20 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Non Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; Lenalidomide; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment-naive DLBCL (Experimental): Treatment-naive high-risk DLBCL patients will be enrolled. R/R2-CHOP were allowed in cycle 1 due to poor physical condition or liver and renal failure caused by lymphoma progression. Patients achieving Complete Remission (CR) or Partial Remission (PR) after 2 cycles will receive another 2 cycles. Patients achieving CR or PR after 4 cycles will finish 6 cycles. Patients achieving CR after 6 cycles with double-hit/triple-hit/double-expression/median to high risk aaIPI will undergo Autologous Stem Cell Transplantation (ASCT). Other patients will be administered rituximab for another 2 cycles and then turn to follow-up. After completion of study treatment, patients are followed up every 3 months for 2 years, and then every 6 months for another 3 years. Patients achieving Stable Disease (SD) or PD (Progression Disease) after 2 or 4 cycles will quit the study. After 6 cycles, patients achieving SD or PD will quit the study and patients achieving PR will receive second-line therapy.
  Interventions: Drug: Zanubrutinib; Drug: Lenalidomide; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone (or equivalent)

INTERVENTIONS:
Drug: Zanubrutinib — 160 mg capsules administered by mouth twice daily (21-day cycles).
Drug: Lenalidomide — 25 mg capsules administered by mouth once daily on Day 1 to Day 10 of each cycle (21-day cycles)
Drug: Rituximab — 375 mg/m2 administered intravenously once on Day 1 of each cycle (21-day cycles)
Drug: Cyclophosphamide — 750 mg/m2 administered intravenously once on Day 1 of each cycle (21-day cycles)
Drug: Doxorubicin — 50 mg/m2 administered intravenously once on Day 1 of each cycle (21-day cycles)
Drug: Vincristine — 1.4 mg/m2 administered intravenously once on Day 1 of each cycle (21-day cycles)
Drug: Prednisone (or equivalent) — 40 mg/m2 capsules administered by mouth once daily on Day 1 to Day 5 of each cycle

SUMMARY:
This study is a multi-center, open-label, single-arm, non-randomized phase II clinical study in order to evaluate the safety and efficacy of zanubrutinib, lenalidomide plus R-CHOP (ZR2-CHOP) as the first-line therapy for treatment-naive high-risk diffuse large B-cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed and previously untreated Diffuse Large B-cell Lymphoma (DLBCL) with median to high risk (including but not limited to double/triple-hit, double expression and median-to-high risk aaIPI).
2. Male or female patients above 18 years old.
3. No prior exposure to treatment except a limited-field radiotherapy, short-term use of glucocorticoid =<25mg/day prednisone equivalent (must discontinue prior to day 1 of cycle 1) and/or cyclophosphamide due to an urgent lymphoma-related clinical situation (e.g. epidural spinal cord compression, superior vena caval syndrome and etc.).
4. At least one measurable disease, as defined as radiographically apparent disease with the longest axis >=1.5cm.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤3 (Patients with ECOG PS 3 should only be included if investigators deem that decline of status due to lymphoma and is reversible).
6. Serum bilirubin <1.5 Upper Limit of Normal (ULN), other than gilbert syndrome (defined as unconjugated bilirubin >80%); Aspartate transaminase (AST) and Alanine aminotransferase (ALT) ≤3 ULN or <5 ULN (if abnormality due to lymphoma).
7. Enough reserve function of bone marrow, regarded as absolute neutrophil count (ANC) > 1.0×109/L and Platelets > 75 ×109/L except that abnormality is due to lymphoma involvement in the bone marrow and felt reversible by investigators.
8. Creatinine clearance rate (Ccr) ≥30 ml / min calculated by Cockcroft-Gault formula.
9. Patients must give consent to transfusions of blood products.
10. Able to take aspirin (100mg) or alternative therapy daily as prophylactic anticoagulation.
11. With life expectancy more than 3 months.
12. All study participants must give consent to follow-up. Patients are fully aware of disease they have and sign informed consent on their own in order to join this study and receive treatment and follow-up.

Exclusion Criteria:

1. Any serious medical condition including but not limited to uncontrolled hypertension, uncontrolled congestive heart failure within past 6 months prior to screening (class 3 [moderate] or class 4 [severe] cardiac disease as defined by the New York Heart Association Functional Classification), uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), left ventricular ejection fraction (LVEF) less than 55%, renal failure, active infection, history of invasive fungal infection, moderate to severe hepatic disease (Child Pugh class B or C), active hemorrhage, laboratory abnormality, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form; patients with history of cardiac arrhythmias should have cardiac evaluation and clearance.
2. Pregnant or lactating females.
3. Known hypersensitivity to lenalidomide or thalidomide, Bruton's Tyrosine Kinase (BTK) inhibitor, rituximab, vincristine, doxorubicin, cyclophosphamide, or prednisone.
4. Patients with active hepatitis B infection (HBV-DNA detectable) and active hepatitis C infection; patients with other acquired or congenital immunodeficiency disease, including but not limited to human immunodeficiency virus (HIV) infection.
5. All patients with central nervous system involvement with lymphoma; patients with primary mediastinal large B cell lymphoma; patients with Richter Syndrome (aggressive DLBCL transformed from indolent CLL).
6. Patients diagnosed as other malignancy except lymphoma, not including:

   Patients received curable treatment and no occurrence of active malignancy more than 5 years prior to study entry; successfully treated basal cell carcinoma without disease symptoms (except melanoma); successfully treated "in situ" cervix carcinoma.
7. Significant neuropathy (grade 2 or grade 1 with pain) within 14 days prior to enrollment.
8. Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis not due to lymphoma.
9. Patients with active pulmonary embolism or deep vein thrombosis (diagnosed within 30 days of study enrollment).
10. Patients with severe bradycardia (heart rate < 40 beats per minute [bpm], hypotension, light-headedness, syncope).
11. Major surgery within 3 weeks of study entry, or wound that is not healed from prior surgery or trauma.
12. History of stroke or intracranial hemorrhage within 6 months prior to study entry.
13. Requires anticoagulation with warfarin or equivalent vitamin K antagonists.
14. Requires chronic treatment with strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors.
15. Vaccinated with live, attenuated vaccines within 4 weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate after six cycles of ZR2-CHOP | at the end of 6 cycles(each cycle is 21 days)
  Complete response rate will be assessed by (18)F-fluorodeoxyglucose (FDG) positron emission tomography (PET/CT) according to 2014 Lugano Criteria.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) two years follow-up | At 2 years
  PFS was defined as the duration from the date of randomization to the date of progression, relapse from CR, or death, whichever occurred first. Responses were based on 2014 Lugano Criteria.
Overall survival (OS) two years follow-up | At 2 years
  Overall survival was defined as the duration from the date of randomization to the date of the participant's death. Median Overall Survival was estimated by using the Kaplan-Meier method.
Circulating tumor Deoxyribonucleic Acid (ctDNA) clearance rate | Baseline (At initial start), at the end of 2,4 ,6 cycles(each cycle is 21 days)
  ctDNA will be measured at baseline and after 2, 4, 6 cycles of ZR2-CHOP
Overall response rate after six cycles of ZR2-CHOP | at the end of 6 cycles(each cycle is 21 days)
  Overall response rate will be assessed by FDG-PET/CT or CT scan according to 2014 Lugano Criteria.
Overall response rate after two, four cycles of ZR2-CHOP | at the end of 2,4 cycles(each cycle is 21 days)
  Overall response rate will be assessed by FDG-PET/CT according to 2014 Lugano Criteria.
Complete response rate after two, four cycles of ZR2-CHOP | at the end of 2,4 cycles(each cycle is 21 days)
  Overall response rate will be assessed by FDG-PET/CT according to 2014 Lugano Criteria.
Incidence of adverse events | At 2 years
  Toxicities will be summarized by grade and by their relationship to treatment according to CTCAE (version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, Phd, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - Department of Haematology, the First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjin, Jiangsu
  - First affiliation hospital of nanjing medical university, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xia Y, Miao Y, Qian S, Zhang R, Qin S, Xie X, Li B, Sha Y, Tang H, Jin H, Cao L, Xu W, Fan L, Li J, Shi W, Zhu H. Zanubrutinib, lenalidomide and rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone as initial treatment in non-germinal center B-cell diffuse large B-cell lymphoma: a multi-center phase 2 study by Jiangsu Cooperative Lymphoma Group (JCLG). BMC Med. 2025 Oct 24;23(1):583. doi: 10.1186/s12916-025-04418-y. PMID 41136989